CLINICAL TRIAL: NCT02657330
Title: A Phase 1A/1B Study of SBP-101 in Previously Treated Subjects With Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Study of SBP-101 in Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Panbela Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-SBP-101-01
Record Dates: First submitted 2015-12-22; First posted 2016-01-15 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Pancreatic Cancer; Ductal Adenocarcinoma of the Pancreas
Keywords: Locally Advanced; Metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBP-101 (Experimental): SBP-101 is administered as a subcutaneous injection once daily, Monday through Friday for 3 weeks (total of 15 doses) followed by a 5-week rest period (3 weeks on, 5 weeks off = 1 treatment cycle). Dose escalation in phase 1a will continue until the maximum tolerated dose is determined.
  Interventions: Drug: SBP-101

INTERVENTIONS:
Drug: SBP-101 — Subcutaneous drug, escalating dose cohorts
  Other Names: diethyl dihydroxyhomospermine; [(HO)2-DEHSPM]

SUMMARY:
This phase 1 first-in-human study evaluates safety and tolerability of SBP-101 in subjects with previously treated pancreatic ductal adenocarcinoma and will identify the maximum tolerated dose (MTD). In addition, this study will also assess the pharmacokinetic (PK) profile and preliminary efficacy of SBP-101.

DETAILED DESCRIPTION:
This first-in-human study of SBP-101 will be conducted in two phases: dose escalation and expansion. The dose escalation phase of the study is to evaluate the safety, tolerability and PK profile of SBP-101 in subjects with previously treated locally advanced or metastatic pancreatic ductal adenocarcinoma. Up to 48 subjects may be enrolled in dose escalation. The expansion phase of the study will consist of 24 additional subjects who will receive the maximum tolerated dose of SBP-101 based on data from the dose escalation phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic pancreatic ductal adenocarcinoma. Patients with acinar cell carcinoma may also be included.
* Measurable disease on CT or MRI scan by RECIST criteria (required for Phase 1b only).
* ECOG Performance Status 0 or 1.
* Received and failed, or were intolerant to, at least 1 prior systemic therapy for locally advanced or metastatic pancreatic ductal adenocarcinoma.
* Adult, at least 18 years of age, male or female
* Females of child-bearing potential must have a negative serum pregnancy test within 14 days prior to start of study treatment and must use an adequate method of contraception during the study. All sexually active males must also use an adequate method of contraception during the study.
* Adequate bone marrow, hepatic, renal and coagulation function as defined by the following: Absolute neutrophil count ≥1.5 x 10^9/L, Hemoglobin ≥9.0 g/dL (90 g/L), Platelets ≥100 x 10^9/L, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN) (if no hepatic metastases). If hepatic tumor involvement, AST and ALT ≤5 x ULN, Bilirubin ≤1.5 x ULN, Prothrombin time (PT) / international normalized ratio (INR) ≤1.5 x ULN, Calculated creatinine clearance >50 mL/min using the Cockcroft and Gault equation
* QTc interval ≤ 470 msec at Baseline
* Willing and able to provide written informed consent: voluntary agreement to participate in the study following disclosure of risks and procedures required, including possibility of onset of exocrine pancreatic insufficiency with subsequent requirement for life-long pancreatic enzyme replacement

Exclusion Criteria:

* Evidence of severe or uncontrolled systemic disease or any concurrent condition that, in the opinion of the Investigator or Medical Monitor, makes it undesirable for the subject to participate in the study or that would jeopardize compliance with the protocol. Subjects with pre-existing well-controlled diabetes are not excluded.
* Medical or psychiatric conditions that compromise the subject's ability to give informed consent or to complete the protocol or a history of non-compliance
* Presence of islet-cell or pancreatic neuroendocrine tumor or mixed adenocarcinoma-neuroendocrine carcinoma
* Have symptomatic central nervous system (CNS) malignancy or metastasis. Screening of asymptomatic subjects without history of CNS metastases is not required.
* Serum albumin <30 g/L (3.0 g/dL)
* Glycosylated hemoglobin (Hgb A1C) > 8.0%
* Life expectancy <16 weeks
* Presence of known active bacterial, fungal, or viral infection requiring systemic therapy
* Known infection with human immunodeficiency virus (HIV), hepatitis B or C
* Presence of interstitial lung disease, pulmonary fibrosis, or pulmonary hypersensitivity reaction
* Myocardial infarction within the last 12 months, severe/unstable angina, symptomatic congestive heart failure, New York Heart Association (NYHA) class III or IV
* Maldigestion/malabsorption syndrome pre-dating the diagnosis of pancreatic cancer.
* Known, existing coagulopathy or receiving anticoagulants
* Pregnant or lactating
* Major surgery within 4 weeks of the start of study treatment, without complete recovery
* Participation in any other clinical investigation within 4 weeks of receiving the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of SBP-101 | Up to 18 months following the first dose of treatment

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | Up to 30 months following the first dose of treatment
Tumor response will be evaluated based on Response Evaluation Criteria in Solid Tumors (RECIST) definitions | Every 8 weeks during treatment assessed up to 30 months
Area under the plasma concentration versus time curve (AUC) | Days 1 and 18 of Cycle 1 (each cycle is 8 weeks)
Peak plasma concentration (Cmax) | Days 1 and 18 of Cycle 1 (each cycle is 8 weeks)
Plasma drug half-life | Days 1 and 18 of Cycle 1 (each cycle is 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Gagnon, MD, Study Director — Panbela Therapeutics, Inc.
Locations (4):
- United States (2):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
- Australia (2):
  - Ashford Cancer Centre, Kurralta Park, South Australia
  - Austin Hospital, Heidelberg, Victoria